CLINICAL TRIAL: NCT03884036
Title: Effect of Vitamin D in Burn Patients: A Randomized Clinical Trial
Brief Title: Effect of Vitamin D in Burn Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hangang Sacred Heart Hospital (Other)
Collaborators: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Hee Yeong Kim, Assistant Professor, Hangang Sacred Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2019-003
Record Dates: First submitted 2019-03-13; First posted 2019-03-21 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Burn Surgery
MeSH Terms: interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D group (Active Comparator): Vitamin D 200,000 IU (1 cc) IM
  Interventions: Biological: Vitamin D
- Control group (Placebo Comparator): Normal saline 1 cc IM
  Interventions: Biological: Vitamin D

INTERVENTIONS:
Biological: Vitamin D — Vitamine D

SUMMARY:
The purpose of this study is to evaluate pre-operative vitamin D levels in patients with burn injuries and evaluate the effect of vitamin D on postoperative complications and duration of hospitalization.

DETAILED DESCRIPTION:
Vitamin D deficiency often occurs in burn patients, which may include longer hospitalization and respiratory and cardiac complications.

The purpose of this study is to evaluate pre-operative vitamin D levels in patients with burn injuries and evaluate the effect of vitamin D on postoperative complications and duration of hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* vitamin D <30 ng/ml
* patients undergoing burn surgery

Exclusion Criteria:

* age < 18 years old
* hypercalcemia
* renal disease
* cardiac disease ( EF<40%, MI, angina)
* respiratory disease (ARDS, pneumonia)
* intubated patients
* electrical burn

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2019-07-18 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative complications | Within postoperative 1 month
  Infection, cardiovascular complication, gastrointestinal complication, respiratory complication, renal complication, and death

SECONDARY OUTCOMES:
Vitamin D level | Within postoperative 14 days
  Serum 25-hydroxy vitamin D level

OTHER OUTCOMES:
Hospital stay | Time from operation to discharge (approximately within 1 month)
  Length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Young-Kug Kim, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Hangang Sacred Heart Hospital, Seoul, South Korea